CLINICAL TRIAL: NCT05545410
Title: Optimization of Thoracic Aortic MRI Acquisition Sequences for the Quantification of Diagnostic-assisting Biomarkers (SEQUOIA)
Brief Title: Optimization of Thoracic Aortic MRI Acquisition Sequences for the Quantification of Diagnostic-assisting Biomarkers
Acronym: SEQUOIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211541
Record Dates: First submitted 2022-08-03; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: thoracic aorta; MRI; acquisition calibration; biomarkers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Other)
  Interventions: Other: MRI calibration

INTERVENTIONS:
Other: MRI calibration — Non-injected thoracic aorta MRI calibration

SUMMARY:
The main objective is to optimize MRI acquisition and image post-processing protocols in order to define the best compromise between short scan time and image quality (contrast between different tissues, spatial and temporal resolutions) high enough to accurately measure morphologic, hemodynamic and structural aortic biomarkers.

DETAILED DESCRIPTION:
This Magnetic Resonance imaging study of the thoracic aorta aims to: 1- enhance patient comfort during the examination, shorten appointment waiting times and overall reduce MRI cost, and 2- provide a reliable diagnosis and risk assessment of aorta-related diseases occurring in hypertension, obesity or diabetes but also throughout normal aging.

The impact of MRI acquisition innovations on the measurement of biomarkers that are extracted from image post-processing software and therein on disease characterization (normal values, severity thresholds, etc.) must be systematically reevaluated. More specifically, the investigators design image acquisition and automated image processing methods to reduce operator variability. This study will optimize thoracic aortic MRI acquisition sequences for the quantification of diagnostic-assisting biomarkers in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 20 and 35 or between 50 and 70 (limits included)
* BMI < 30 kg/m²
* Asymptomatic subject
* Having given informed, free and written consent
* Affiliated to a French social security scheme or entitled

Exclusion Criteria:

* Contraindication to MRI (claustrophobia, presence of a metallic foreign body)
* Pregnant or breastfeeding woman
* Known cardiac pathology
* Personal cardiovascular history
* Person deprived of liberty by court decision or benefiting from legal protection (under guardianship or curatorship)
* Abuse of alcohol or narcotics
* Subject under AME
* Participation in another interventional research involving the human person or being in the exclusion period at the end of a previous research involving the human person

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Parametric measurement of thoracic aorta values of normal subjects | 24 months
  Thoracic aorta values measured by MRI

SECONDARY OUTCOMES:
Quantitative fibrosis within the aortic wall (%) | 24 months
Quantitative fat within the aortic wall (%) | 24 months
Quantitative periaortic fat (g and g/m², when indexed to BSA) | 24 months
ROC metrics will be used to compare the various sequences (%) | 24 months
Quantitative flow values within the different aortic segments and the main branches (mL) | 24 months
Correlation coefficients will be estimated to assess the associations between novel and conventional biomarkers | 24 months
Intra and inter-reproductibility of aortic measures will be assessed (intra-class correlation coefficients) | 24 months
Intra and inter-reproductibility of aortic measures will be assessed (Bland and Altman metrics) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raluca PAIS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal